CLINICAL TRIAL: NCT01062659
Title: Characterization of Cellular Immune Responses in the Liver in Patients With Chronic Hepatitis C Virus Infection
Brief Title: Cellular Immune Responses in the Liver in Chronic Hepatitis C (CHC) Patients
Status: Withdrawn | Type: Observational
Why Stopped: Lack of funding
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Dietmar M. Klass, Dr. med., University of Ulm
Other Study IDs: TCell
Record Dates: First submitted 2010-02-03; First posted 2010-02-04 (Estimated); Last update posted 2014-04-01 (Estimated); Status verified 2014-03

CONDITIONS: Hepatitis C, Chronic; Liver Diseases; Virus Diseases
Keywords: HCV; hepatitis C virus; CHC; chronic hepatitis c; interferon; ribavirin; Hepatitis, Viral, Human; Anti-Infective Agents; peginterferon alfa-2a; peginterferon alfa-2b
MeSH Terms: conditions — Hepatitis C, Chronic; Liver Diseases; Virus Diseases; Hepatitis C; Hepatitis, Viral, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- chronic Hepatitis C: Patients with chronic Hepatitis C (CHC) Genotype 1-4 who are naive to antiviral treatment

SUMMARY:
In order to persist in the liver, HCV has numerous nonspecific and specific strategies to overcome the immunity of the host. The crucial step in the establishment of viral persistence and chronic hepatitis is the avoidance of specific antiviral cellular immune response in the liver. Treatment with pegylated interferon alpha (IFNα) in combination with ribavirin (RBV) is the standard therapy for chronic hepatitis C is. The response to IFNα / RBV therapy depends on the effective cellular antiviral immune response in the liver. The understanding of the interaction between HCV and cellular immune response is important for the effective use of existing diagnostic techniques, the Individual control and adjustment of the current therapeutic approaches and the development of future therapeutic and immunization strategies. In this study, the investigators want to investigate cellular Immune responses in the liver of HCV infected patients and characterize the influence of these immune responses to the response to IFNα / RBV therapy.

ELIGIBILITY:
Inclusion Criteria:

* proven chronic hepatitis C
* aged between 18 and 65
* willingness to give written informed consent to the study protocol

Exclusion Criteria:

* history of having received any IFN, PEG-IFN or RBV
* not eligible for antiviral treatment with peginterferon and ribavirin by standard of care

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patient with established chronic hepatitis C presented to the liver unit of the outpatient clinic how are eligible to antiviral therapy.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-02; Primary Completion 2012-12 (Estimated); Study Completion 2013-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Dietmar M Klass, MD, Principal Investigator — University of Ulm
Locations (1):
- University Hospital Ulm, Ulm, Germany